CLINICAL TRIAL: NCT03457077
Title: Neural and Mobile Assessment OF Behavior Change Among Problem Drinkers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Northwell Health (Other)
Responsible Party: Principal Investigator, Nasir Naqvi, research psychiatrist, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 7390
Record Dates: First submitted 2018-03-01; First posted 2018-03-07 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-07

CONDITIONS: Alcohol Use Disorder
Keywords: brief intervention; fMRI
MeSH Terms: conditions — Alcoholism | interventions — Crisis Intervention

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief Intervention (Experimental): Participants will receive a brief intervention at week 0
  Interventions: Behavioral: Brief intervention
- Delayed Intervention (Other): Participants will receive a brief intervention at 6 months
  Interventions: Behavioral: Brief intervention

INTERVENTIONS:
Behavioral: Brief intervention — A brief motivational intervention with feedback about drinking levels compared to norms

SUMMARY:
This study will examine the neural mechanisms underlying both spontaneous behavior change and behavior change in response to a brief intervention among problem drinkers.

DETAILED DESCRIPTION:
Although problem drinkers (PD) are a less severe, highly prevalent sub-type of alcohol use disorder (AUD) who are more likely to undergo reductions in alcohol use, compared to more severe AUD, the underlying mechanisms that maintain PD, as well as the mechanisms that underlie both spontaneous and treatment- related behavior change in this population, are not well understood. This proposal takes a lab to life approach by combining functional neuroimaging (fMRI), ecological momentary assessment (EMA), and brief interventions (BI) in non-treatment seeking PD to test whether heightened incentive salience (reactivity) to alcohol cues and impaired ability to regulate cue-induce craving are the mechanisms that characterize PD, and play a role in behavior change vs. persistence of behavior. Identifying these mechanisms is critical for testing and understanding treatments and uncovering who is most likely to respond to interventions.

ELIGIBILITY:
Inclusion Criteria (Problem Drinkers):

* Age 21-55
* English language fluency
* Over the last 28 days ,Have an average weekly consumption of greater than 14 standard drinks for women, and greater than 24 standard drinks for men.
* Current DSM-V mild or moderate alcohol use disorder (AUD) diagnosis
* Own a smartphone with data plan

Inclusion Criteria (Healthy Controls):

* Age 21-55
* English language fluency
* Have an average weekly consumption of less than </=14 standard drinks for women and less than/equal to 24 standard drinks for men and up to 2 heavy drinking days (>4/5 standard drinks for a woman/man)
* No lifetime diagnosis of AUD
* owns smartphone with a data plan

Exclusion Criteria:

* Past or current severe AUD as defined by DSM- V
* Currently seeking treatment or attempting to stop drinking
* Past or current alcohol withdrawal symptoms
* Current DSM-V diagnosis of substance use disorder (other than nicotine or caffeine).
* Regular use (more than 1-2 times weekly) of recreational drugs.
* Psychotic Disorder or Bipolar disorder
* Severe depression (Patient Health Questionnaire score > 19) or anxiety (Beck Anxiety Inventory > 25)
* Substantial risk of suicide or violence
* MRI contraindications (e.g., metallic implants, pacemaker, weight > 350 lbs, waist > 55")
* Hearing impaired/hearing aids, unable to read newspaper at arm's length with corrective
* Objective cognitive impairment
* Current or recent (evidence of disease x 5 years) non-skin neoplastic disease or melanoma. - Active hepatic disease (not a history of hepatitis) or primary renal disease requiring dialysis, primary untreated endocrine diseases, e.g., Cushing's disease or primary hypothalamic failure or insulin dependent diabetes (Type I or II). Well-treated hypothyroidism will not be excluded.
* Pregnant, lactating (participation allowed 3 months after ceasing lactation), or currently intending to become pregnant
* Any history of ECT
* Brain disorder such as stroke, tumor, infection, epilepsy, multiple sclerosis, degenerative diseases, head injury (LOC > 5 minutes), mental retardation
* Diagnosed learning disability, dyslexia, or ADHD
* For women: Current pregnancy or intention to be pregnant in the near future

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 164 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Drinking | 6 months
  Heavy drinking days

CONTACTS AND LOCATIONS:
Overall Officials: Nasir Naqvi, MD, PhD, Principal Investigator — Columbia University
Locations (1):
- NYPInstitute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No